CLINICAL TRIAL: NCT06410950
Title: Exploring Muscle Proprieties in COPD: a Non-invasive Evaluation of Respiratory and Limb Muscle Mechanics Using Myotonometry.
Brief Title: Mechanical Muscle Proprieties in Patient with COPD
Status: Completed | Type: Observational
Sponsor: Spitalul Clinic de Boli Infecțioase și Pneumoftiziologie Dr. Victor Babeș Timișoara (Other Government)
Responsible Party: Principal Investigator, Crisan Alexandru Florian, Principal Investigator, Spitalul Clinic de Boli Infecțioase și Pneumoftiziologie Dr. Victor Babeș Timișoara
Other Study IDs: 3654/04
Record Dates: First submitted 2024-04-22; First posted 2024-05-13 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-09

CONDITIONS: Copd; Muscle Weakness; Muscle Weakness Condition
Keywords: COPD; Muscle tone; Muscle stiffness; Muscle mechanical proprieties
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Muscle Weakness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- COPD subjects: Individuals diagnosed with COPD based on GOLD spirometry criteria (post-bronchodilator FEV1/FVC ratio < 0.70).
  Stable COPD with no exacerbations requiring hospitalization in the past six months.
  Age range: 45-75 years old.
  Interventions: Diagnostic Test: MyotonPRO Assessment of Muscle Biomechanical Properties
- Healthy subjects: Individuals with no history of chronic respiratory disease or recent infections.
  Normal lung function on spirometry (post-bronchodilator FEV1/FVC ratio > 0.70). Age range: 40-75 years old.
  Interventions: Diagnostic Test: MyotonPRO Assessment of Muscle Biomechanical Properties

INTERVENTIONS:
Diagnostic Test: MyotonPRO Assessment of Muscle Biomechanical Properties — Muscle assessments will be conducted using the MyotonPRO (Myoton AS., Tallinn, Estonia) digital palpation device. Measurement patterns and subject data will be uploaded to the device via computer. Each evaluation will be performed bilaterally.
  Subjects' muscle measurement points will be marked prior to assessment. The physiotherapist will position the device perpendicular to the muscle body and apply downward pressure (18N). Pressure should be maintained until the device's probe light changes from red to green. Five measurement pulses will then be applied. Each pulse lasts 15 ms with an 8 ms interval between pulses.
  The SENIAM sensor location guide will be used to determine the approximate motor point for MyotonPRO measurements.

SUMMARY:
This study aims to determine if patients with Chronic Obstructive Pulmonary Disease (COPD) exhibit altered muscle properties (specifically changes in tone and stiffness) in both their respiratory muscles and skeletal muscles when compared to healthy individuals. The study will utilize the Myotonometer, a non-invasive device, to assess these properties.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) leads to progressive airflow limitation and respiratory muscle dysfunction, contributing to exercise intolerance and reduced quality of life. While existing methods evaluate overall lung function, the assessment of specific respiratory muscle properties remains challenging. Myotonometry offers a non-invasive technique to quantify muscle tone and stiffness, potentially providing insights into respiratory and skeletal muscle mechanics in COPD. This study aims to explore differences in the mechanical properties of both superficial respiratory and skeletal muscles in patients with COPD compared to healthy controls using myotonometry. Investigators hypothesize that COPD patients will exhibit altered mechanical properties (e.g., increased stiffness and tone) in both superficial respiratory and skeletal muscles compared to healthy controls.

ELIGIBILITY:
Inclusion criteria for the COPD group:

Diagnosis of COPD: Confirmed diagnosis of COPD based on GOLD spirometry criteria:

Post-bronchodilator FEV1/FVC ratio < 0.70 Documented history of respiratory symptoms (e.g., dyspnea, cough, sputum production) Stable COPD: No COPD exacerbations requiring hospitalization in the past 6 months.

Smoking History: Current or former smoker with a documented smoking history of at least 10 pack-years (cumulative cigarette consumption).

Age: 45-75 years old. Ability to Understand and Follow Instructions: Mentally competent and able to understand the study procedures, risks, and benefits, providing written informed consent.

Exclusion criteria for the COPD group:

Other respiratory disease than COPD. Severe COPD exacerbation: anyone with a COPD exacerbation requiring hospitalization within the last six months.

Conditions limiting chest wall movement: severe kyphosis, ankylosing spondylitis, or similar conditions that significantly impact the ability to expand the chest wall and perform respiratory muscle assessments.

Muscular or neuromuscular disorders: primary muscular diseases (e.g., muscular dystrophy) or neuromuscular disorders affecting muscle function (e.g., Parkinson's, multiple sclerosis).

Recent Surgery or Trauma: Significant surgery or trauma within the past three months that might affect muscle function or the ability to perform assessments.

Uncontrolled comorbidities: severe, uncontrolled medical conditions that could significantly impact muscle function or confound the study results (e.g., uncontrolled heart failure, advanced renal disease).

Inclusion criteria for the healthy control group:

No History of Respiratory Disease: free from any current or past respiratory diagnoses, including asthma, chronic bronchitis, or recurrent respiratory infections.

Normal lung function: spirometry testing will confirm normal lung function with a post-bronchodilator FEV1/FVC ratio > 0.70 and no evidence of airflow obstruction.

No significant chronic conditions: free from any major chronic medical conditions that could impact muscle function or confound the results (e.g., uncontrolled diabetes, heart failure, advanced liver disease).

Age: 45-75 years old Ability to understand and follow instructions: mentally competent and able to understand the study procedures, risks, and benefits, providing written informed consent.

No recent infections: free from any recent respiratory or other infections within the past 4 weeks.

Non-smoker or minimal smoking history: non-smokers or have a very minimal smoking history (less than 10 pack-years)

Exclusion criteria for the healthy control group:

Recent respiratory infection: anyone with a current respiratory tract infection (viral or bacterial) within the past four weeks.

Mild respiratory symptoms: Even mild, persistent respiratory symptoms (chronic cough, sputum production) within the past 4 weeks.

Conditions limiting chest wall movement: severe kyphosis, ankylosing spondylitis, or similar conditions that significantly impact the ability to expand the chest wall and perform respiratory muscle assessments.

Muscular or neuromuscular disorders: primary muscular diseases (e.g., muscular dystrophy) or neuromuscular disorders affecting muscle function (e.g., Parkinson's, multiple sclerosis).

Recent Surgery or Trauma: Significant surgery or trauma within the past three months that might affect muscle function or the ability to perform assessments.

Uncontrolled comorbidities: severe, uncontrolled medical conditions that could significantly impact muscle function or confound the study results (e.g., uncontrolled heart failure, advanced renal disease).

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with COPD and healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Semispinalis capitis state of tension | Baseline
  To assess the tension of the semispinalis capitis (SC), participants will lie in a supine position on the treatment table. The physiotherapist will identify the measurement point using a pencil. This point will be located approximately two finger widths lateral to the spinous process of the C7 vertebra and slightly inferior to the occiput (base of the skull). The device will be held vertically and a consistent downward pressure of 18 Newtons (N) will be applied to the muscle belly. Once the indicator light on the probe transitions from red to green, pressure will be maintained while the MyotonPRO delivers five stimulation pulses. The following will be assessed:
  Tone or state of tension: F - Natural Oscillation Frequency [Hz].
Semispinalis capitis biomechanical properties | Baseline
  To assess the biomechanical properties of the semispinalis capitis (SC), participants will lie in a supine position on the treatment table. The physiotherapist will identify the measurement point using a pencil. This point will be located approximately two finger widths lateral to the spinous process of the C7 vertebra and slightly inferior to the occiput (base of the skull). The device will be held vertically and a consistent downward pressure of 18 Newtons (N) will be applied to the muscle belly. Once the indicator light on the probe transitions from red to green, pressure will be maintained while the MyotonPRO delivers five stimulation pulses. The following will be assessed:
  Biomechanical properties: S-Dynamic Stiffness [N/m].
Semispinalis capitis viscoelastic properties | Baseline
  To assess the viscoelastic properties of the semispinalis capitis (SC), participants will lie in a supine position on the treatment table. The physiotherapist will identify the measurement point using a pencil. This point will be located approximately two finger widths lateral to the spinous process of the C7 vertebra and slightly inferior to the occiput (base of the skull). The device will be held vertically and a consistent downward pressure of 18 Newtons (N) will be applied to the muscle belly. Once the indicator light on the probe transitions from red to green, pressure will be maintained while the MyotonPRO delivers five stimulation pulses. The following will be assessed:
  Viscoelastic properties: R-Mechanical Stress Relaxation Time [ms].
Sternocleidomastoideus (SCM) state of tension | Baseline
  To assess the tension of the sternocleidomastoideus (SCM), participants will lie supine on the treatment table. The evaluator will locate the midpoint on a line between the mastoid process (behind the ear) and the clavicle (collarbone), marking this point with a pencil. The device will be held vertically and a consistent downward pressure of 18 Newtons (N) will be applied to the muscle belly. Once the indicator light on the probe transitions from red to green, pressure will be maintained while the MyotonPRO delivers five stimulation pulses. The following will be assessed:
  Tone or state of tension: F - Natural Oscillation Frequency [Hz].
Sternocleidomastoideus (SCM) biomechanical properties | Baseline
  To assess the biomechanical properties of the sternocleidomastoideus (SCM), participants will lie supine on the treatment table. The evaluator will locate the midpoint on a line between the mastoid process (behind the ear) and the clavicle (collarbone), marking this point with a pencil. The device will be held vertically and a consistent downward pressure of 18 Newtons (N) will be applied to the muscle belly. Once the indicator light on the probe transitions from red to green, pressure will be maintained while the MyotonPRO delivers five stimulation pulses. The following will be assessed:
  Biomechanical properties: S-Dynamic Stiffness [N/m].
Sternocleidomastoideus (SCM) viscoelastic properties | Baseline
  To assess the viscoelastic properties of the sternocleidomastoideus (SCM), participants will lie supine on the treatment table. The evaluator will locate the midpoint on a line between the mastoid process (behind the ear) and the clavicle (collarbone), marking this point with a pencil. The device will be held vertically and a consistent downward pressure of 18 Newtons (N) will be applied to the muscle belly. Once the indicator light on the probe transitions from red to green, pressure will be maintained while the MyotonPRO delivers five stimulation pulses. The following will be assessed:
  Viscoelastic properties: R-Mechanical Stress Relaxation Time [ms].
Trapezius state of tension | Baseline
  To assess the tension of the trapezius, participants will sit upright in a chair with good back support. Their hips should touch the back of the chair, feet flat on the floor, and hands resting comfortably in their lap. Shoulders will be relaxed, and knees and hips bent at a 90-degree angle. The upper trapezius measurement point is midway between the C7 vertebra (prominent at the base of the neck) and the acromion (the bony tip of the shoulder). The following will be assessed:
  Tone or state of tension: F - Natural Oscillation Frequency [Hz].
Trapezius biomechanical properties | Baseline
  To assess the biomechanical properties of the trapezius, participants will sit upright in a chair with good back support. Their hips should touch the back of the chair, feet flat on the floor, and hands resting comfortably in their lap. Shoulders will be relaxed, and knees and hips bent at a 90-degree angle. The upper trapezius measurement point is midway between the C7 vertebra (prominent at the base of the neck) and the acromion (the bony tip of the shoulder). The following will be assessed:
  Biomechanical properties: S-Dynamic Stiffness [N/m].
Trapezius viscoelastic properties | Baseline
  To assess the viscoelastic properties of the trapezius, participants will sit upright in a chair with good back support. Their hips should touch the back of the chair, feet flat on the floor, and hands resting comfortably in their lap. Shoulders will be relaxed, and knees and hips bent at a 90-degree angle. The upper trapezius measurement point is midway between the C7 vertebra (prominent at the base of the neck) and the acromion (the bony tip of the shoulder). The following will be assessed:
  Viscoelastic properties: R-Mechanical Stress Relaxation Time [ms].
Deltoid state of tension | Baseline
  To assess deltoid tension, participants will lie in the supine position. The physiotherapist will locate the measurement point using a pencil. This point will be roughly halfway down the muscle, centered between the lateral aspect of the acromion process (bony point of the shoulder) and the insertion point on the deltoid tuberosity (bumpy area near the midpoint of the upper arm bone). The following will be assessed:
  Tone or state of tension: F - Natural Oscillation Frequency [Hz].
Deltoid biomechanical properties | Baseline
  To assess the biomechanical properties of the deltoid muscle, participants will lie in the supine position. The physiotherapist will locate the measurement point using a pencil. This point will be roughly halfway down the muscle, centered between the lateral aspect of the acromion process (bony point of the shoulder) and the insertion point on the deltoid tuberosity (bumpy area near the midpoint of the upper arm bone). The following will be assessed:
  Biomechanical properties: S-Dynamic Stiffness [N/m].
Deltoid viscoelastic properties | Baseline
  To assess deltoid viscoelastic properties, participants will lie in the supine position. The physiotherapist will locate the measurement point using a pencil. This point will be roughly halfway down the muscle, centered between the lateral aspect of the acromion process (bony point of the shoulder) and the insertion point on the deltoid tuberosity (bumpy area near the midpoint of the upper arm bone). The following will be assessed:
  Viscoelastic properties: R-Mechanical Stress Relaxation Time [ms].
Biceps brahii state of tension | Baseline
  To assess biceps brachii tension, participants will lie supine on the treatment table with their arms at their sides and palms facing upwards. The physiotherapist will locate the measurement point on the front of the upper arm, approximately midway between the shoulder and elbow crease. Using a pencil, they will mark this point. The following will be assessed:
  Tone or state of tension: F - Natural Oscillation Frequency [Hz].
Biceps brahii biomechanical properties | Baseline
  To assess the biomechanical properties of biceps brachii, participants will lie supine on the treatment table with their arms at their sides and palms facing upwards. The physiotherapist will locate the measurement point on the front of the upper arm, approximately midway between the shoulder and elbow crease. Using a pencil, they will mark this point. The following will be assessed:
  Biomechanical properties: S-Dynamic Stiffness [N/m].
Biceps brahii viscoelastic properties | Baseline
  To assess the biceps brachii viscoelastic properties, participants will lie supine on the treatment table with their arms at their sides and palms facing upwards. The physiotherapist will locate the measurement point on the front of the upper arm, approximately midway between the shoulder and elbow crease. Using a pencil, they will mark this point. The following will be assessed:
  Viscoelastic properties: R-Mechanical Stress Relaxation Time [ms].
Brachioradialis state of tension | Baseline
  To assess brachioradialis tension, participants will lie supine on the treatment table with their arms at their sides and palms facing upwards. The physiotherapist will locate the measurement point on the front of the upper arm, approximately midway between the shoulder and elbow crease. Using a pencil, they will mark this point. The device will be held vertically and a steady downward pressure of 18 Newtons (N) will be applied directly over the marked point. Once the indicator light on the probe transitions from red to green, pressure will be maintained while the MyotonPRO delivers five stimulation pulses. The following will be assessed:
  Tone or state of tension: F - Natural Oscillation Frequency [Hz].
Brachioradialis biomechanical properties | Baseline
  To assess the biomechanical properties of brachioradialis, participants will lie supine on the treatment table with their arms at their sides and palms facing upwards. The physiotherapist will locate the measurement point on the front of the upper arm, approximately midway between the shoulder and elbow crease. Using a pencil, they will mark this point. The device will be held vertically and a steady downward pressure of 18 Newtons (N) will be applied directly over the marked point. Once the indicator light on the probe transitions from red to green, pressure will be maintained while the MyotonPRO delivers five stimulation pulses. The following will be assessed:
  Biomechanical properties: S-Dynamic Stiffness [N/m].
Brachioradialis viscoelastic properties | Baseline
  To assess brachioradialis viscoelastic properties, participants will lie supine on the treatment table with their arms at their sides and palms facing upwards. The physiotherapist will locate the measurement point on the front of the upper arm, approximately midway between the shoulder and elbow crease. Using a pencil, they will mark this point. The device will be held vertically and a steady downward pressure of 18 Newtons (N) will be applied directly over the marked point. Once the indicator light on the probe transitions from red to green, pressure will be maintained while the MyotonPRO delivers five stimulation pulses. The following will be assessed:
  Viscoelastic properties: R-Mechanical Stress Relaxation Time [ms].
Rectus femoris state of tension | Baseline
  To assess rectus femoris tension, participants will lie supine on a treatment table. The physiotherapist will locate the measurement point along the front of the thigh, approximately halfway between the anterior superior iliac spine (hip bone) and the top of the patella (kneecap). A pencil will be used to mark this point. The device will be held vertically, and a steady downward pressure of 18 Newtons (N) will be applied directly over the marked point. Once the indicator light on the probe transitions from red to green, pressure will be maintained while the MyotonPRO delivers five stimulation pulses. The following will be assessed:
  Tone or state of tension: F - Natural Oscillation Frequency [Hz].
Rectus femoris biomechanical properties | Baseline
  To assess the biomechanical properties of the rectus femoris, participants will lie supine on a treatment table. The physiotherapist will locate the measurement point along the front of the thigh, approximately halfway between the anterior superior iliac spine (hip bone) and the top of the patella (kneecap). A pencil will be used to mark this point. The device will be held vertically, and a steady downward pressure of 18 Newtons (N) will be applied directly over the marked point. Once the indicator light on the probe transitions from red to green, pressure will be maintained while the MyotonPRO delivers five stimulation pulses. The following will be assessed:
  Biomechanical properties: S-Dynamic Stiffness [N/m].
Rectus femoris viscoelastic properties | Baseline
  To assess rectus femoris viscoelastic properties, participants will lie supine on a treatment table. The physiotherapist will locate the measurement point along the front of the thigh, approximately halfway between the anterior superior iliac spine (hip bone) and the top of the patella (kneecap). A pencil will be used to mark this point. The device will be held vertically, and a steady downward pressure of 18 Newtons (N) will be applied directly over the marked point. Once the indicator light on the probe transitions from red to green, pressure will be maintained while the MyotonPRO delivers five stimulation pulses. The following will be assessed:
  TViscoelastic properties: R-Mechanical Stress Relaxation Time [ms].
Vastus medialis state of tension | Baseline
  To assess vastus medialis tension, participants will lie in a supine position on the treatment table with their legs extended. The physiotherapist will locate the measurement point on the inner thigh, approximately one hand-width above the superior-medial border of the patella (kneecap). This point should align with the visible bulge of the vastus medialis muscle. A pencil will be used to mark this point. The following will be assessed:
  Tone or state of tension: F - Natural Oscillation Frequency [Hz].
Vastus medialis biomechanical properties | Baseline
  To assess vastus medialis biomechanical properties, participants will lie in a supine position on the treatment table with their legs extended. The physiotherapist will locate the measurement point on the inner thigh, approximately one hand-width above the superior-medial border of the patella (kneecap). This point should align with the visible bulge of the vastus medialis muscle.A pencil will be used to mark this point. The following will be assessed:
  Biomechanical properties: S-Dynamic Stiffness [N/m].
Vastus medialis viscoelastic properties | Baseline
  To assess vastus medialis viscoelastic properties, participants will lie in a supine position on the treatment table with their legs extended. The physiotherapist will locate the measurement point on the inner thigh, approximately one hand-width above the superior-medial border of the patella (kneecap). This point should align with the visible bulge of the vastus medialis muscle.A pencil will be used to mark this point. The following will be assessed:
  Viscoelastic properties: R-Mechanical Stress Relaxation Time [ms].
Vastus lateralis state of tension | Baseline
  To assess vastus lateralis tension, participants will lie in a supine position on the treatment table with their leg extended. The physiotherapist will locate the measurement point on the outer thigh, approximately one hand-width above the superior-lateral border of the patella (kneecap). This point should align with the pronounced bulge of the vastus lateralis muscle. The following will be assessed:
  Tone or state of tension: F - Natural Oscillation Frequency [Hz].
Vastus lateralis biomechanical properties | Baseline
  To assess vastus lateralis biomechanical properties, participants will lie in a supine position on the treatment table with their leg extended. The physiotherapist will locate the measurement point on the outer thigh, approximately one hand-width above the superior-lateral border of the patella (kneecap). This point should align with the pronounced bulge of the vastus lateralis muscle. The following will be assessed:
  Biomechanical properties: S-Dynamic Stiffness [N/m].
Vastus lateralis viscoelastic properties | Baseline
  To assess vastus lateralis viscoelastic properties, participants will lie in a supine position on the treatment table with their leg extended. The physiotherapist will locate the measurement point on the outer thigh, approximately one hand-width above the superior-lateral border of the patella (kneecap). This point should align with the pronounced bulge of the vastus lateralis muscle. The following will be assessed:
  Viscoelastic properties: R-Mechanical Stress Relaxation Time [ms].
Tibialis anterior state of tension | Baseline
  To assess tibialis anterior tension, participants will sit comfortably in a chair with their feet flat on the floor. The physiotherapist will locate the measurement point on the front of the lower leg, approximately one-third of the distance between the knee and the ankle. This point typically aligns with the most prominent bulge of the tibialis anterior muscle. The following will be assessed:
  Tone or state of tension: F - Natural Oscillation Frequency [Hz].
Tibialis anterior biomechanical properties | Baseline
  To assess tibialis anterior biomechanical properties, participants will sit comfortably in a chair with their feet flat on the floor. The physiotherapist will locate the measurement point on the front of the lower leg, approximately one-third of the distance between the knee and the ankle. This point typically aligns with the most prominent bulge of the tibialis anterior muscle. The following will be assessed:
  Biomechanical properties: S-Dynamic Stiffness [N/m].
Tibialis anterior viscoelastic properties | Baseline
  To assess tibialis anterior viscoelastic properties, participants will sit comfortably in a chair with their feet flat on the floor. The physiotherapist will locate the measurement point on the front of the lower leg, approximately one-third of the distance between the knee and the ankle. This point typically aligns with the most prominent bulge of the tibialis anterior muscle. The following will be assessed:
  Viscoelastic properties: R-Mechanical Stress Relaxation Time [ms].

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru Crișan, PhD, Principal Investigator — Spitalul Clinic de Boli Infecțioase și Pneumoftiziologie Dr. Victor Babeș Timișoara
Locations (1):
- Spitalul de Boli Infectioase si Pneumoftiziologie Victor Babes, Timișoara, Timiș County, Romania